CLINICAL TRIAL: NCT02607332
Title: A Trial of Paclitaxel in Patients With Metastatic or Advanced Gastrointestinal Stromal Tumors (GIST) After Failure to Imatinib and Sunitinib
Brief Title: Paclitaxel in Patients With Metastatic or Advanced Gastrointestinal Stromal Tumors (GIST) After Failure to Imatinib and Sunitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1501
Record Dates: First submitted 2015-11-12; First posted 2015-11-18 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: single-center; prospective; single-arm; open-label; phase II
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel (Experimental): paclitaxel 80mg/m2/day on a Cycle1Day1, Cycle1Day8,Cycle1Day15 off 1 week schedule
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel

SUMMARY:
With discovery of KIT mutations and the advent of KIT tyrosine kinase inhibitor imatinib (GlivecTM, Novartis), there has been substantial improvement in overall survival in patients with advanced and/or metastatic gastrointestinal tumors (GIST). Recently, sunitinib (SuteneTM, Pfizer) showed activity as second-line therapy in GIST patients after failure with imatinib. However, virtually all patients will eventually progress or become intolerable after the first-line imatinib and the second-line sunitinib.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older
* Histologically confirmed metastatic and/or advanced GIST with CD117(cluster of differentiation 117)(+), DOG-1(+), or mutation in KIT or PDGFRα gene(Platelet Derived Growth Factor Receptor)
* Failed (progressed and/or intolerable) after prior treatments for GIST, including at least both imatinib and sunitinib .
* Eastern Cooperative Oncology Group performance status of 0~2
* Resolution of all toxic effects of prior treatments to grade 0 or 1 by NCI-Common Toxicity Criteria for Adverse Effects version 3.0
* At least one measurable lesion as defined by Response Evaluation Criteria In Solid Tumors version 1.0
* Adequate bone marrow, hepatic, renal, and other organ functions

  * Neutrophil > 1,500/mm3
  * Platelet > 100,000/mm3
  * Hemoglobin > 8.0 g/dL
  * Total bilirubin < 1.5 x upper limit of normal (ULN)
  * Aspartate aminotransferase /Alanine transferase< 2.5 x ULN (or < 5 x ULM in case of liver metastases)
  * Creatinine < 1.5 x ULN
* Life expectancy > 12 weeks
* Washout period of previous TKIs(Tyrosine Kinase Inhibitor) or chemotherapy for more than 4 times the half life.
* Provision of a signed written informed consent

Exclusion Criteria:

* Women of child-bearing potential who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control.
* have the presence of cardiac disease,including a myocardial infarction within 6 months prior to study entry,Clinically significant cardiac disease (New York Heart Association, Class III or IV) or severe unstable angina pectoris, stroke or transient ischemic attack, Arrhythmia in need of treatment
* Uncontrolled infection
* Diabetes mellitus (insulin dependent or independent disease, requiring chronic medication) with signs of clinically significant peripheral vascular disease.
* Acute and chronic liver disease and all chronic liver impairment.(Patients with stable and chronic viral hepatitis are eligible are acceptable)
* Uncontrolled gastrointestinal toxicities with toxicity greater than NCI Common Toxicity Criteria for Adverse Effects grade 2
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality.
* The patient experienced any bleeding episode considered life-threatening, or any grade 3 or 4 bleeding event.
* Major surgery ≤ 28 days prior to starting study drug or who have not recovered from side effects of such therapy.
* Known diagnosis of HIV infection .
* History of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Patients with brain metastases as assessed by radiologic imaging
* Alcohol or substance abuse disorder.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Disease control rate | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea